CLINICAL TRIAL: NCT06289205
Title: Comparison of Peroperative Methotrexate Infusion With Postoperative Intra Silicon Oil Methotrexate Injections for Prevention of Proliferative Vitreoretinopathy Development After Vitrectomy for Rhegmatogenous Retinal Detachment Repair.
Brief Title: "Comparing Methotrexate Usage Techniques to Prevent Proliferative Vitreoretinopaty After Retinal Detachment Vitrectomy"
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Ahmad Zeeshan Jamil, Professor of Ophthalmology, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 60/IRB/SLMC/SWL
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Proliferative Vitreoretinopathy
Keywords: Methotrexate; Retinal detachment; Vitrectomy; Proliferative Vitreoretinopathy
MeSH Terms: conditions — Vitreoretinopathy, Proliferative; Retinal Detachment | interventions — Methotrexate; Antimetabolites

STUDY DESIGN:
Intervention Model Description: Using lottery methods patients will be divided into two groups with 60 subjects in each group. Group 1 will be regarded as control group and per operative methotrexate infusion will be used by mixing 75 mg of methotrexate into one litre of BSS solution. Group 2 will be regarded as the study group and will receive 500 µg of intra-silicon oil methotrexate at the end of the surgery and then at 1st, 2nd, 3rd , 4th and 6th post operative weeks.
Who Masked: Participant
Masking Description: This will be a single-blind study in which the subjects will be unaware of the intervention. Blinding will be maintained by ensuring that subjects are unaware of the dosing regimens they are receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 will be regarded as control group and per operative methotrexate infusion will be used by mixing 75 mg of methotrexate into one litre of BSS solution.
  Interventions: Drug: Methotrexate
- Group 2 (Experimental): Group 2 will be regarded as the study group and will receive 500 µg of intra-silicon oil methotrexate at the end of the surgery and then at 1st, 2nd, 3rd , 4th and 6th post operative weeks.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Methotrexate will be utilised in two different ways to prevent development of proliferative vitreoretinopathy after vitrectomy for rhegmatogenous retinal detachment
  Other Names: Antimetabolite

SUMMARY:
This clinical trial, involving participants with rhegmatogenous retinal detachment, aims to compare Methotrexate Usage Techniques in preventing Proliferative Vitreoretinopathy (PVR) after vitrectomy. The study will evaluate the development of PVR, retinal detachment recurrence, and improvement in visual acuity. Participants will undergo retinal detachment surgery using the vitrectomy technique and will be divided into two groups. One group will receive Methotrexate infusion during surgery, while the other will receive repeated Methotrexate injections post-surgery. The researcher will analyze and compare outcomes between the two groups.

DETAILED DESCRIPTION:
This interventional trial will be conducted at the Sahiwal Teaching Hospital, Sahiwal and Ali Fatima Teaching Hospital Lahore from March 2024 to May 2025. The study will follow the guidelines of the Declaration of Helsinki. The study protocol will be approved by institutional review boards of respective hospitals. Written informed consent will be taken from all the subjects. The first subject will be recruited in March 2024 and the last subject will be recruited in February 2025. Three more months will be required to complete the final follow-up of the last subject.

The study will include rhegmatogenous retinal detachments patients of both sexes between 20 and 70 years of age.

Exclusion criteria will include the presence of proliferative vitreoretinopathy grade C, previous retinal detachment surgery in the same eye, penetrating ocular trauma, intraocular foreign bodies, and pregnant and lactating women.

A detailed history of the patients' presenting complaints, duration of symptoms, and risk factors for retinal detachment will be gathered. Comprehensive ocular examination, including visual acuity, intraocular pressure, and examination of the anterior and posterior segments, will be performed. The extent of retinal detachment, location of retinal breaks, and presence of PVR will be documented.

Sampling method will be simple random sampling. Using lottery methods patients will be divided into two groups with 60 subjects in each group. Group 1 will be regarded as control group and per operative methotrexate infusion will be used by mixing 75 mg of methotrexate into one litre of BSS solution. Group 2 will be regarded as the study group and will receive 500 µg of intra-silicon oil methotrexate at the end of the surgery and then at 1st, 2nd, 3rd , 4th and 6th post operative weeks.

This will be a single-blind study in which the subjects will be unaware of the intervention. Blinding will be maintained by ensuring that subjects are unaware of the dosing regimens they are receiving.

Standard pars plana vitrectomy will be performed by two surgeons, one surgeon at Sahiwal Teaching Hospital Sahiwal and other surgeon at Ali Fatima Teaching Hospital Lahore. Silicon oil will be used as post operative tamponade in all subjects. A combination of steroid and antibiotic eye drops will be administered eight times per day during the first postoperative week. The dosing will be tapered off during the next three weeks. Patients will be instructed to adopt the appropriate posture according to the location of retinal breaks.

Follow-up will be performed every week for three months. The development of PVR, occurrence of retinal detachment, intraocular pressure, and visual acuity will be noted. The posterior segment will be examined with the help of a superfield lens and wide-field contact lens for the development of PVR and occurrence of retinal detachment.

The primary outcomes will be the development of PVR and the recurrence of retinal detachment. All patients will be followed up until the development of one of the primary outcomes or completion of 3 month follow, whichever occurs earlier.

Improvement in visual acuity will be secondary outcome of the study. Final visual acuity will be measured at completion of 3 month follow up or meeting the primary outcome, whichever is earlier.

All information will be collected using a specially designed proforma and entered into SPSS version 26. Qualitative variables, such as sex, PVR development, recurrence of retinal detachment, and improvement in visual acuity, will be presented as frequencies and percentages. Quantitative variables, such as age and intraocular pressure, are presented as mean and standard deviation.

In this prospective study we shall investigate the differences in the development of proliferative vitreoretinopathy (PVR) between two distinct groups. Additionally, we shall compare the difference in the occurrence of re-detachment of the retina between these groups. Furthermore, we shall compare the improvement in visual acuity at the final follow-up visit between the two groups. As the variables involved will be qualitative (frequency of eyes with development of PVR, Frequency of eyes with retinal re-detachment, and frequency of eyes with improved visual acuity), Pearson's chi-square test will be used to carry out the statistical analysis. Statistical significance will set at P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Rhegmatogenous Retinal Detachment

Exclusion Criteria:

* Presence of proliferative vitreoretinopathy grade C, previous retinal detachment surgery in the same eye, penetrating ocular trauma, Presence of intraocular foreign bodies, previous glaucoma filtration surgery, allergy to methotrexate, and pregnant and lactating women.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Development of Proliferative Vitreoretinopathy (PVR) | Within three months of Vitrectomy surgery
  Clinically evident PVR membrane formation
Recurrence of Retinal Detachment | Within three months of Vitrectomy surgery
  Re detachment of retina after retinal detachment repair surgery by vitrectomy

SECONDARY OUTCOMES:
Visual Acuity Improvement | Final visual acuity will be measured at completion of 3 month follow up or meeting the primary outcome, whichever is earlier.
  Improvement in visual acuity after retinal detachment repair by vitrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Z Jamil, FCPS,FRCS, Principal Investigator — Sahiwal Medical College, Sahiwal, Pakistan
Locations (1):
- Sahiwal Medical College & Teaching Hospital, Sahiwal, Pakistan, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
For sharing IPD, ethica approval will be sought from institutional review board. Privacy of participants will be maintained and unique identifiers will be used to track the individual participants. Participants history, surgical records and follow up visits will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting six months after publishing, data will become available for one year.
Access Criteria: Access will be granted for legitimate and scientifically sound research purposes that align with the objectives of the original study. Access will be contingent upon the ability of the requesting researchers to adhere to rigorous data security and privacy measures to safeguard participant confidentiality. Researchers should provide information on their intent to publish the results of their analysis, promoting transparency and accountability in the use of shared data. Requesting researchers must agree to and sign a Data Use Agreement (DUA) outlining the terms and conditions of data use, including restrictions, publication policies, and compliance with ethical standards.

REFERENCES:
- [Result] Nagpal M, Chaudhary P, Wachasundar S, Eltayib A, Raihan A. Management of recurrent rhegmatogenous retinal detachment. Indian J Ophthalmol. 2018 Dec;66(12):1763-1771. doi: 10.4103/ijo.IJO_1212_18. PMID 30451176
- [Result] El Baha S, Leila M, Amr A, Lolah MMA. Anatomical and Functional Outcomes of Vitrectomy with/without Intravitreal Methotrexate Infusion for Management of Proliferative Vitreoretinopathy Secondary to Rhegmatogenous Retinal Detachment. J Ophthalmol. 2021 Jul 20;2021:3648134. doi: 10.1155/2021/3648134. eCollection 2021. PMID 34336257
- [Result] Jahangir S, Jahangir T, Ali MH, Lateef Q, Hamza U, Tayyab H. Use of Intravitreal Methotrexate Infusion in Complicated Retinal Detachment for Prevention of Proliferative Vitreoretinopathy in a Pilot Study. Cureus. 2021 Aug 25;13(8):e17439. doi: 10.7759/cureus.17439. eCollection 2021 Aug. PMID 34462712

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT06289205/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT06289205/ICF_001.pdf